CLINICAL TRIAL: NCT06919848
Title: Oncolytic Virus H101 Combined With Lenvatinib Plus Toripalimab Compared With FOLFOX in Patients With Advanced Biliary Tract Cancer (OPTIONS-06): a Multicenter, Randomized, Phase 2 Study
Brief Title: Oncolytic Virus H101 Combined With Lenvatinib Plus Toripalimab Compared With FOLFOX in Patients With Advanced Biliary Tract Cancer (OPTIONS-06)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIONS-06
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Biliary Tract Cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — lenvatinib; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H101+ lenvatinib+Toripalimab (Experimental): H101 combined with lenvatinib plus Toripalimab
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 ); Drug: Lenvatinib; Drug: H101
- FOLFOX (Active Comparator): FOLFOX chemotherapy
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) — Toripalimab will be administered by IV, 240 mg on day 1 of each 21 day cycle until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Arms: H101+ lenvatinib+Toripalimab
Drug: Lenvatinib — Lenvatinib will be administered (bodyweight ≥ 60 kg, 12 mg; < 60 kg, 8 mg) orally daily until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Arms: H101+ lenvatinib+Toripalimab
Drug: H101 — H101 will be percutaneously injected into tumor on day 1 of every 21-day cycle. Lenvatinib plus Toripalizumab will be administered 1-3 days after H101 injection.
  Arms: H101+ lenvatinib+Toripalimab
Drug: FOLFOX — FOLFOX chemotherapy was administered intravenously every 2 weeks for a maximum of 12 cycles (oxaliplatin 85 mg/m², leucovorin, 400 mg/m2, fluorouracil 400 mg/m² [bolus], and fluorouracil 2400 mg/m² as a 46-h continuous intravenous infusion
  Arms: FOLFOX

SUMMARY:
This study will evaluate the efficacy and safety of Oncolytic virus H101 combined with lenvatinib plus Toripalimab compared with FOLFOX in patients with advanced biliary tract cancer (BTC) who have progressed after first-line treatment.

DETAILED DESCRIPTION:
The participants will be randomized in a 1:1 ratio to one of the two treatment arms: Arm A (experimental arm): H101 + lenvatinib + Toripalimab; Arm B (control arm): FOLFOX

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Participants must have unresectable or metastatic histologically or cytologically confirmed biliary tract cancer.
* Participants must have failed 1 line of systemic regimens for advanced cholangiocarcinoma due to disease progression or toxicity.
* At least one measurable site of disease as defined by RECIST criteria with spiral CT scan or MRI.
* Performance status (PS) ≤ 2 (ECOG scale).
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥75 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior treatment with oncolytic virus.
* Prior treatment with Lenvatinib or other targeted therapy.
* RFA and resection administered less than 4 weeks prior to study treatment start.
* Radiotherapy administered less than 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to: a) history of interstitial lung disease b) Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection) c) known acute or chronic pancreatitis d) active tuberculosis e) any other active infection (viral, fungal or bacterial) requiring systemic therapy f) history of allogeneic tissue/solid organ transplant g) diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment. h) Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study. i) Live vaccine within 30 days prior to the first dose of treatment or during study treatment. j) History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Prior therapy with an anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 42 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD).
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Time to Response (TTR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  TTR is defined as the time from the start of treatment until the first objective observation of a response (either partial response, PR, or complete response, CR), provided that the response is subsequently confirmed.
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.
Translational study | max 42 months
  Proportion of different immune cell types in tumors based on RNA sequencing between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No